CLINICAL TRIAL: NCT00939406
Title: A Multi-center Prospective Randomized Phase II Clinical Trial to Evaluate Safety and Efficacy of Hyalospine® in Lumbar Laminectomy or Laminotomy
Brief Title: Clinical Trial to Evaluate Safety and Efficacy of Hyalospine® in Lumbar Laminectomy or Laminotomy
Acronym: Hyalospine
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: AO Clinical Investigation and Publishing Documentation (Other)
Responsible Party: Sponsor
Organization: AO Innovation Translation Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Hyalospine
Record Dates: First submitted 2009-07-14; First posted 2009-07-15 (Estimated); Last update posted 2012-12-20 (Estimated); Status verified 2012-12

CONDITIONS: Degenerative Spinal Stenosis; Disk Herniation
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Control group consists of subjects randomized to the control arm who will receive lumbar decompression surgery (laminotomy or laminectomy) alone
- Hyalospine (Experimental): Intervention group consists of subjects randomized to the treatment arm who will receive lumbar decompression surgery (laminotomy or laminectomy) and HyaloSpine.
  Interventions: Device: Hyalospine

INTERVENTIONS:
Device: Hyalospine — Intervention group consists of subjects randomized to the treatment arm who will receive lumbar decompression surgery (laminotomy or laminectomy) and HyaloSpine.
  Arms: Hyalospine

SUMMARY:
The aim of this Phase II trial is to evaluate safety and efficacy of Hyalospine in patients undergoing lumbar laminectomy or laminotomy for degenerative spinal stenosis or disk herniation. The device is used as an adjunct in lumbar spine surgery to prevent post- surgical fibrosis and adhesions, and improve patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for elective single- or two-level lumbar laminectomy or laminotomy procedure for treatment of spinal stenosis and/or disk herniation.
* Subjects who have failed conservative care for at least 6 weeks.

Exclusion Criteria:

* Contraindication to MRI
* Instrumented fusion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2009-11; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Rate of adverse events | 6 months
Extent of epidural fibrosis | 12 months

SECONDARY OUTCOMES:
differences in pain, neurological status, neurological symptoms, function, quality of life, patient satisfaction, immunologic and clinical laboratory results | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Paul Pavlov, MD, Principal Investigator — Sint Maartenskliniek, Nijmegen, The Netherlands
Locations (3):
- Zentrum für Wirbelsäulenchirurgie und Neurotraumatologie, BG Unfallklinik Frankfurt/Main, Frankfurt, Germany
- Sint Maartenskliniek, Nijmegen, The Netherlands, Woerden, Netherlands
- Klinik Sonnehof, Bern, Canton of Bern, Switzerland